CLINICAL TRIAL: NCT01297699
Title: Clinical Trial Phase III, Parallel Group, Randomized, Placebo-controlled, Double-blind, Multicenter Study to Evaluate the Efficacy and Safety of Tocilizumab Administration in Patients With Moderate-to-severe or Sight-threatening Graves' Ophthalmopathy (GO), That Had Not Responded Adequately to Treatment With Intravenous Corticoid Pulses.
Brief Title: Tocilizumab Treatment in Graves´ Ophthalmopathy (Graves´ Orbitopathy or Thyroid Eye Disease)
Acronym: GRC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Collaborators: Fundación Ramón Domínguez (Other)
Responsible Party: Principal Investigator, Dr. Juan Jesus Gomez-Reino Carnota, MD, PhD, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GRC-TCL-2010-01; 2010-023841-31 (EudraCT Number)
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Thyroid Associated Ophthalmopathies; Graves´ Ophthalmopathy; Thyroid Eye Disease
Keywords: Graves´ orbitopathy; Graves´ ophthalmopathy; Thyroid eye disease; Thyroid-associated ophthalmopathy; Tocilizumab; EUGOGO; CAS
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — tocilizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tocilizumab (Experimental)
  Interventions: Drug: Tocilizumab (RoActemra®)
- Sterile 0.9% Sodium Chloride (Placebo Comparator)
  Interventions: Drug: Sterile 0.9% Sodium Chloride

INTERVENTIONS:
Drug: Tocilizumab (RoActemra®) — Single intravenous infusion of tocilizumab (8 mg/kg); every 4 weeks during 16 weeks.
  Arms: Tocilizumab
Drug: Sterile 0.9% Sodium Chloride — Single intravenous dip infusion of a sterile 0.9% sodium chloride, every four weeks during 16 weeks.
  Arms: Sterile 0.9% Sodium Chloride

SUMMARY:
The purpose is to investigate tocilizumab administration in patients with moderately to severely or sight-threatening GO (Graves' ophthalmopathy) without response to treatment with corticoid intravenous pulses. Currently, these patients only have surgery as therapeutic alternative.

The principal aim of this study is to evaluate efficacy and safety of tocilizumab treatment in order to provide a better alternative to surgery for this patients.

DETAILED DESCRIPTION:
Thyroid orbitopathy or Graves´orbitopathy (GO) is manifested for inflammation of the orbital and periorbital soft tissues. Ten percent of patients with GO will have long-term serious eye problems.

The cause of the GO is complex. Autoreactive T cells recognize an autoantigen, the TSH receptor present in the orbit and thyroid follicular cell, secrete cytokines (IL-6), which stimulate the fibroblasts to synthesize glycosaminoglycan, which draws liquid produce periorbital edema and muscle, causing exophthalmos.

This approach suggests that inhibition of IL-6 can be an effective treatment for this problem on the basis that tocilizumab specifically binds to the receptors of the IL-6, both soluble and membrane-bound. Tocilizumab has been shown to inhibit signaling mediated for IL-6Rm IL-6Rs.

ELIGIBILITY:
Principal Inclusion Criteria:

Patients diagnosed GO with CAS ≥ 4 and an index of severity, according EUGOGO guidelines, 1. moderately to severely or 2. sight-threatening GO, after receiving corticosteroid pulse treatment due to:

* Poor response to intravenous corticosteroid pulses Or
* Recurrence of the GO, after treatment with intravenous corticosteroids

Exclusion Criteria:

* Orbital decompression surgery needed immediately
* Active smoker
* Patients who could need treatment with radioactive iodine or thyroidectomy during the study
* Pregnant patient or patient who is planning to become pregnant during the study
* History of chronic recurrent or active infection
* History of intestinal ulceration or diverticulitis
* Patients with a history of chronic liver disease or liver disorders: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) above 5 times upper limit of normal (ULN)
* History of HIV, hepatitis C or hepatitis B Positive
* Neutrophil count < 0.5 × 109/L or a platelet count < 50×103/μL
* Simultaneous use or contraindications to the use of immunosuppressive agents
* A treatment with another investigational drug within four weeks of selection or five half-lives of study drug
* Cardiovascular or cerebrovascular disease clinically significant
* Uncontrolled diabetes mellitus
* Use of corticosteroids during four weeks before to inclusion period
* History of reactions or anaphylactic allergic severe human monoclonal antibodies, humanized or murine
* Uncontrolled pathologies, whose exacerbations are treated with corticosteroids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-03; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Drug efficacy will be established as a decrease in CAS (clinical activity score) by 2 or more points in a scale of 10. | It will be measured before treatment (week -4 / 0), after treatment (week 16) and after the end of the follow-up (week 40).

SECONDARY OUTCOMES:
Clinical response of patients who respond to treatment with tocilizumab | It will be analyzed before treatment (week -4 / 0), after treatment (week 16) and once to follow up (week 40).
Evaluate the patients quality of life associated with tocilizumab treatment, using SF-36 | It will be analyzed before treatment (week -4 / 0), after treatment (week 16) and once to follow up (week 40).
Determine time to recurrence during follow-up period | It is measured on a weeks-time scale assessed by the physician during patient follow-up visits.
Safety as adverse events reported | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Juan Jesús Gómez-Reino Carnota, MD, PhD, Study Chair — Hospital Clínico de Santiago; Jóse V. Pérez Moreiras, MD, PhD, Principal Investigator — Centro Oftalmológico Moreiras
Locations (9):
- Spain (9):
  - Hospital Clínico de Santiago, Santiago de Compostela, A Coruña
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Centro Oftalmológico Moreiras, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario La Fe, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza